CLINICAL TRIAL: NCT04629716
Title: Medical Marijuana Use and Driving Performance: A Test of Psychomotor Function in Adults 50 and Older
Brief Title: Reactions of Older Adults Driving After Cannabis Exposure
Acronym: ROADACE
Status: Completed | Type: Observational
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Nicole Ennis, Associate Professor, Florida State University
Other Study IDs: STUDY00001659
Record Dates: First submitted 2020-11-10; First posted 2020-11-16 (Actual); Results first posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Chronic Pain
Keywords: medical marijuana; older adults; chronic pain
MeSH Terms: conditions — Chronic Pain | interventions — Medical Marijuana

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention: The intervention group will be comprised of adults 50 and older who report severe or chronic pain, are newly registered for the Medical Marijuana Registry in the State of Florida, have no prior history of medical marijuana use, can communicate in English, and are willing and able to complete study procedures. The control group will be age, sex, and race matched. The primary study outcome is simulated driving performance (i.e. errors in response time, attention, and executive functioning tasks that predict on-road performance). Secondary outcomes include adverse effects.
  Interventions: Other: Medical Cannabis
- Control: The control group will be comprised of adults 50 and older who report severe or chronic pain, have no prior history of medical marijuana use, can communicate in English, and are willing and able to complete study procedures. The control group will be age, sex, and race matched. The primary study outcome is simulated driving performance (i.e. errors in response time, attention, and executive functioning tasks that predict on-road performance). Secondary outcomes include adverse effects.

INTERVENTIONS:
Other: Medical Cannabis — Medical marijuana is defined by Florida state statue 381.986 as all parts of any plant of the genus Cannabis, whether growing or not; the seeds thereof; the resin extracted from any part of the plant; and every compound, manufacture, salt, derivative, mixture, or preparation of the plant or its seeds or resin, including low-THC cannabis, which are dispensed from a medical marijuana treatment center for medical use by a qualified patient.
  Other Names: Medical Marijuana
  Groups: Intervention

SUMMARY:
Objective of the Protocol: The primary aim of the current protocol is to examine whether or not habitual use of medical marijuana affects psychomotor functioning operationalized as driving performance. Secondary endpoints will examine whether type of medical marijuana used, frequency, dosage or route of administration is associated with Unwanted effects. The proposed study is a prospective repeated measures experimental study designed to test medical marijuana use as the exposure variable in adults age 50 and older and driving errors in response time, attention, and executive functions as the primary outcome. Secondary outcomes include: Unwanted effects. Participants will complete 3 assessments over a 3 month time period. The 3 assessment time points are: baseline (T1), prior to starting medical marijuana, 1 month post-medical marijuana initiation (T2), and 3 months post-medical marijuana initiation (T3). Electronic Medical Review (EMR) will be conducted at baseline, 1, and 3 months. In addition, potentially confounding disease, treatment, and sociodemographic characteristics will be examined. Data will be collected in a manner that is consistent with transparent reporting as mandated by CONSORT guidelines. Finite mixture modeling and generalized linear modeling accounting for individual and group level outcomes will be used to test the study hypotheses. The investigators propose to enroll 60 adults (n=30 medical marijuana users and n=30 age, race, sex matched controls) ages 50 and older with chronic/severe non-malignant pain, which is the most common diagnosis for medical marijuana users. Primary Endpoint: Thus, the proposed study will test medical marijuana use as the exposure variable in adults age 50 and older and simulated driving performance (e.g. errors in response time, attention, and executive functioning tasks that predict on-road performance) as the primary outcome. Secondary Endpoint: Further, the investigators will explore the association between medical marijuana use and Unwanted effects.

DETAILED DESCRIPTION:
The proposed study is a prospective repeated measures experimental study designed to test medical marijuana use as the exposure variable in adults age 50 and older and driving errors in response time, attention, and executive functions as the primary outcome. Secondary outcomes include: unwanted effects. Participants will complete 3 assessments over a 3-month time period. The 3 assessment time points are: baseline (T1) prior to starting medical marijuana, 1 month post-medical marijuana initiation (T2), and 3 months post-medical marijuana initiation (T3). Electronic Medical Review (EMR) will be conducted at baseline, 1 and 3 months. In addition, potentially confounding disease, treatment, and sociodemographic characteristics will be examined. Data will be collected in a manner that is consistent with transparent reporting as mandated by CONSORT guidelines. Finite mixture modeling and generalized linear modeling accounting for individual and group level outcomes will be used to test the study hypotheses.

Participants will be N=60 adults ages 50 and older who have newly registered with the state of Florida to obtain medical marijuana (n=30) or age, race, sex matched non-marijuana user controls (n=30).

Intervention Group Recruitment. Participants will be recruited from Medical Marijuana Treatment Clinics of Florida's (MMTC) Gainesville location. Recruitment for this study begins pre-medical marijuana exposure. To obtain medical marijuana in the state of Florida there are four steps:

* Step 1: Determine Eligibility: Eligibility for medical marijuana use must be determined by a qualified physician. A patient must first seek treatment from a qualified physician. MMTC has qualified physicians who determine patient eligibility.
* Step 2: Medical Marijuana Registration: Once the MMTC physician determines the patient is eligible for medical marijuana, the physician then inputs the patient's information and the medical marijuana order information into the Medical Marijuana Use Registry. MMTC physicians complete this process during the eligibility appointment. Recruitment for the current project begins at step 2 which is prior to any exposure to medical marijuana. Participants will undergo a brief screen during their visit with the MMTC physician to determine if they meet eligibility criteria (See Eligibility Criteria in Human Study Record 1 per new National Institute of Health (NIH) guidelines). Eligibility screening procedures will be institution review board (IRB)-approved and will not collect any identifying information. Self-report questionnaires will be use to discern eligibility. Eligibility will be confirmed using medical records at enrollment. If MMTC patients meet eligibility criteria, they will be given the opportunity to meet with the study research assistant (RA) to learn more about the project. Participants will be provided a detailed description of the study, and the research assistant will obtain permission to follow up with the patient (by phone or text) in order to track their progress on obtaining their registry identification card.
* Step 3: Medical Marijuana Use Registry Identification Card: Once a physician has input the patient's information into the Medical Marijuana Use Registry (i.e. step 2), the patient is able to apply for a medical marijuana card. This process takes approximately 10-14 days. Participants will be instructed to schedule their baseline study visit prior to obtaining their first dose of medical marijuana. At the baseline appointment the study staff will obtain informed consent and complete the biobehavioral assessment measures, and participants will complete their first drive.
* Step 4: Dispensation of Medical Marijuana: Once the patient receives the medical marijuana card, the patient is then able to fill their first order for medical marijuana at a dispensary. The Medical Marijuana Use Registry will track patients' dose, frequency, type of medical marijuana received, and route of administration. After obtaining their medical marijuana card and filling their first dispensation, the investigators will track patients through MMTC and follow patients for 3 months post medical marijuana initiation.

Control Group Recruitment. Control participants will be age, race, and sex matched adults 50 and older with a diagnosis of chronic or severe pain recruited from the community using flyers/handouts; newspaper/Internet advertisements; in-person lectures and events; and contact via mail, e-mail, and the infrastructure and support of Oak Hammock at the University of Florida (UF), a residential retirement community. The investigators will also phone individuals enrolled in the UF HealthStreet and Clinical and Translational Science Institute's (CTSI) Integrated Data Repository, a database organizing clinical information across UF Health's clinical and research programs.

Attrition is a large concern in an observational trial of this rigor. Within the lab, based on prior experience the investigators anticipate between 15-20% dropout by time point 3. Therefore, the investigators anticipate recruiting 72 participants (62+20%) in order to achieve our goal. However, there are numerous strategies that the investigators have used in the past and will put in place to increase retention.

Test of Aim 1 (Driving Simulator)

Driving Simulator Data will be collected via the kinematic functionality of the high-fidelity driving simulator (e.g. speed in mph, braking, swerving, lateral lane positioning, etc.) and also through observing the performance of the driver via a trained evaluator who will use the playback function of the simulator to scrutinize the errors. The drive will begin with a 5-minute acclimation scenario which is designed to train drivers on aspects of simulator operation and help them adjust to driving in a simulator. The simulator acclimation drive addresses lane keeping on straight and curved roads, braking, changing lanes, use of side and rear-view mirrors, and stopping. After the 5-minute acclimation scenario, the driver will drive the main drive for 10 minutes. Three scripted events will be randomly presented to the drivers to control for learning effects.

* Event 1. To assess response time, during the drive a vehicle is pulling out in front of the driver and the driver's behavior is measured via braking milliseconds (ms) and swerving (standard deviation {SD} of lateral deviation from center lane).
* Event 2. Next, using an established protocol, during the course of the drives four divided attention tasks (being aware of the traffic and surrounding while focusing on critical stimulus) are assessed via a triangle appearing on the screen and the participant needing to press a button (i.e. respond) as soon as they see it (measured in ms and number of omissions and commissions).
* Event 3. Lastly, executive functions are measured by providing the driver with instructions before the drive (i.e. to turn into an onscreen Kentucky Fried Chicken (KFC), pull into a parking bay, and when it is safe to do so, exit the lot and merge into the flow of traffic (measured via visual scanning (yes/no) speed regulation (mph over or under the speed limit), adjustment to stimuli (notice the KFC (yes/no), slow down (mph), signaling (yes/no), vehicle positioning (buffer around the vehicle yes/no), and gap acceptance (narrow or tight via ms)69, 70,121-122. Participants will be scored on number of tasks completed correctly.

Within Subject Analysis. To answer the primary question of this proposal, "Does medical marijuana use affect driving performance?," the investigators will use repeated measures ANOVA. The investigators will examine within subject differences on measures at all 3 time points in order to answer the question of whether medical marijuana impacts response time, divided attention, and executive functions. Using a repeated measures ANOVA, time will serve as the independent variable and continuous measures of driving errors (as defined above) as the outcomes. Power Analysis: The investigators computed the power to detect a medium effect size of 0.5 standard deviations across groups. Assuming a correlation of 0.2 across the repeated measures at three time points, the standard deviation of the average of three measures is 0.683 times the standard deviation of one measure. Therefore, with 30 per group the investigators can detect a difference in this average of 0.5 times the standard deviation of one measure, using a two-sided test with 80% power. The investigators calculated Cohen's d using Dr. Classen's prior work that examined total driving errors and specific errors (lane maintenance) in healthy controls (M=24.08 SD=12.38) and (M=5.78 SD=4.26) versus Parkinson's patients (M=31.99 SD=22.01) and (M=10.23 SD=9.26), which yielded a Cohen's d of .46-.65 (medium effect size)59; therefore, the investigators will be powered to detect this medium effect size.

Between Group Analyses Comparisons between medical marijuana users and control group participants will be examined using independent samples t-test (controlling for unequal variances using Levene's test) or Mann-Whitney U tests if the data are nonparametric in order to rule out change over time as an explanation of findings. No difference is hypothesized between groups at baseline. At time 2 and 3 the control group is hypothesized to have higher average response time, divided attention reaction time, and scores on divided attention tasks completed correctly than medical marijuana users.

Test of Aim 2 (Unwanted Effects) Adverse Effects. In this study, adverse effects are defined as undesired effects that occur when medication is administered. The investigators will use Scripted Prompting, a proactive form of adverse effect capture recognized in the field. This method is designed to elicit adverse effects without biasing the patient; it is a standardized question that allows participants to report important symptoms without being influenced by suggestion. For this study the investigators will ask: "Since initiating medical marijuana, are you having any problems related to use?"

To describe factors associated with adverse effects, the investigators will report the number of adverse effects reported by participants at time points 2 and 3. Unwanted Effects will be defined as both a count variable and a binary variable such that absence or presence of adverse effects will be coded as 0/1 respectively. The investigators will then use Poisson and Logistic regression methods to examine analyze the bivariate association between dosage, frequency of use, route of administration (pills, vape, etc.), and type of product (THC v. CBD). Power Statement: The goal of aim 2 is to examine the strength of the association between factors of medical marijuana use and adverse effects. Currently, the literature does not contain data regarding the strength of the association between medical marijuana use and adverse effects or how dosage, frequency of use, and route of administration are associated with adverse effects. As there may be insufficient power for statistical significance using the proposed analyses above, effect size estimates will be used to examine the strength of the association between variables. With 30 per group, the investigators can detect a difference of 0.73 standard deviations using a two-sided test with 80% power.

Exploratory Aim: Examine factors associated with study feasibility (enrollment and retention) for development of a future R01. The investigators will describe the association between socio-demographic factors (i.e. gender, race, and education) and enrollment and retention in the intervention condition in order to identify ways to improve study feasibility. The investigators will use chi-square for dichotomous variables and Pearson correlations for continuous variables to examine associations between sociodemographic factors and study enrollment (number screened who meet criteria versus number enrolled) and retention (number enrolled versus number completing all 3 time points). This method will allow us to identify candidate predictors of enrollment and attrition to inform the investigative team about strengthening recruitment/retention efforts for specific subgroups.

ELIGIBILITY:
Inclusion Criteria:

* Participant is aged 50 or older
* Participant reports severe and/or chronic pain
* Participant is newly registered to the Medical Marijuana Use Registry in Florida (intervention group only)
* Participant has no prior history with medical marijuana use (intervention group only)

Exclusion Criteria:

* Participant lacks fluency in English
* Participant is unwilling to provide information for follow-up
* Participant plans to leave the area within 3 months
* Participant is unable to provide informed consent due to cognitive impairment
* Participant is unwilling to complete necessary study procedures

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The investigators will recruit 30 patients from Medical Marijuana Treatment Clinics (MMTC) of Gainesville. The intervention group will be comprised of adults 50 and older who report severe or chronic pain, are newly registered for the Medical Marijuana Registry in the State of Florida, have no prior history of medical marijuana use, can communicate in English, and are willing and able to complete study procedures. The control group will be age, sex, and race matched.
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2021-04-23 (Actual); Primary Completion 2023-08-17 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Ennis, PhD, Principal Investigator — Florida State University
Locations (1):
- Smart House at Oak Hammock, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
This data contains medical marijuana status and driving performance outcomes; therefore, it is imperative that we use extensive precautions in protecting the identities of participants. Identifiers will be removed from the data. In order to fully protect the human participants, we will make an evaluation of each data request to ensure that special circumstances do not exist that would permit anyone to deduce the identification of individuals from the remaining data. Based on our evaluation of appropriateness to share data requested, we will make the data and associated documentation available to users under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed.
Supporting Information: Study Protocol
Time Frame: Data will be available six months after Aim 1 and Aim 2 papers have been published
Access Criteria: available to users under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Control
Started (This is Timepoint 1 Baseline) | 23 | 21
Timepoint 2 (This is timepoint 2 approximately one month after initiation of medical marijuana use) | 19 | 19
Completed (This is timepoint 3 approximately 3 months after initiation of medical marijuana use) | 16 | 18
Not Completed | 7 | 3
Not completed — Lost to Follow-up | 7 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 23 | 21 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 11 | 26
  >=65 years | 8 | 10 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.48 (6.42) | 64.24 (6.68) | 62.80 (6.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 11 | 19
  Male | 15 | 10 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 22 | 21 | 43
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 21 | 20 | 41
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 23 | 21 | 44
Center for Epidemiologic Studies Depression ScaleCES-D [Mean (Standard Deviation); unit: units on a scale] — The CES-D is a 20-item self-report questionnaire used to assess depressive symptoms. Each item is rated on a 4-point scale, from 0 (rarely or none of the time) to 3 (most or all of the time).
  0-15: No significant depression 16-19: Mild depression 20-23: Moderate depression 24 or higher: Severe depression
  units on a scale | 16.3 (10.23) | 8.38 (6.06) | 12.52 (9.31)
Mini-Mental State Examination-2; Brief Version (MMSE-2;BV) [Mean (Standard Deviation); unit: units on a scale] — The Mini-Mental State Examination-2; Brief Version is a shorter version of the standard Mini Mental State exam, designed for quick cognitive screening. It yields a total score16. Higher scores are best with those 50 and older expected to score 14 or higher This is a sum scored measure in which you add up the points from each of the four assessed areas: registration, orientation to time, orientation to place, and recall, with each area potentially contributing a maximum of 4 points, resulting in a total possible score of 16 points; a higher score indicates better cognitive function.
  units on a scale | 15.17 (1.15) | 15.43 (0.60) | 15.30 (0.93)
Education [Count of Participants; unit: Participants]
  Less than H.S. | 1 | 0 | 1
  H.S. or GED equivalent | 3 | 2 | 5
  Post H.S. education | 19 | 19 | 38
Income [Count of Participants; unit: Participants]
  Less than 30K USD annual | 5 | 7 | 12
  30,001-60,000 USD annual | 9 | 5 | 14
  60,001 and greater USD annual | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Simulated Driving Performance Task Measuring Divided Attention
Description: Studies of driving performance using driving simulators have been shown to be a valid predictor of on-road driving performance. Driving simulators allow for the systematic presentation of events and the manipulation of variables, which offers experimental control that is impossible on the road. Driving simulators also offer optimal stimulus presentation which allows for analysis of both healthy and impaired drivers under similar conditions. There was a total of 4 divided attention task events presented during the course of the simulated drive. Therefore, scores ranged from 0-4, with 0 indicating poor divided attention (worse outcome) such that all divided attention tasks presented in the simulator was missed and 4 indicating good divided attention (better outcome) such that all divided attention tasks presented in the simulator were completed. Therefore, a higher score indicates better divided attention such that participants attended to more events while driving in the simulator.
Time Frame: 1 month
Population: Primary outcome was analyzed at T2 and each group lost a few participants to follow-up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 19 | 19
units on a scale | 3.42 (0.67) | 2.57 (0.98)

2. Secondary Outcome: Unwanted Effects of Marijuana Use
Description: In this study, adverse effects are defined as undesired effects that occur when the medication is administered. The investigators will use Scripted Prompting, a proactive form of adverse effect capture recognized in the field. This method is designed to elicit adverse effects without biasing the patient; it is a standardized question that allows participant to report important symptoms without being influenced by suggestion. For this study, the investigators will ask: "Since initiating medical marijuana, are you having any problems related to use?"
Time Frame: 1 month
Population: Data available at T2 due to lost to follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 19 | 19
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: Data was collected throughout the course of the study at: Baseline, Timepoint 2 and Timepoint 3 Baseline to timepoint 2 = 1 month Baseline to timepoint 3 = 3 months
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/21
Other Adverse Events (participants affected / at risk) | 0/23 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-10-30): https://cdn.clinicaltrials.gov/large-docs/16/NCT04629716/Prot_SAP_000.pdf
  • Informed Consent Form (2021-04-09): https://cdn.clinicaltrials.gov/large-docs/16/NCT04629716/ICF_001.pdf